CLINICAL TRIAL: NCT05595642
Title: A Phase III, Randomized, Double-Blind, Placebo-Controlled, Multicenter Study to Evaluate the Efficacy and Safety of Astegolimab in Patients With Chronic Obstructive Pulmonary Disease
Brief Title: A Study to Evaluate Astegolimab in Participants With Chronic Obstructive Pulmonary Disease
Acronym: ARNASA
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GB44332; 2022-502234-70-00 (EU CTIS Number)
Record Dates: First submitted 2022-10-24; First posted 2022-10-27 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — astegolimab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Astegolimab SC Q2W (Experimental): Participants will receive subcutaneous (SC) astegolimab every 2 weeks (Q2W)
  Interventions: Drug: Astegolimab
- Astegolimab SC Q4W (Experimental): Participants will receive alternating SC astegolimab and placebo Q2W, thus receiving SC astegolimab Q4W.
  Interventions: Drug: Astegolimab
- Placebo SC Q2W (Placebo Comparator): Participants will receive SC placebo Q2W
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Astegolimab — Participants will receive SC astegolimab Q2W or Q4W
  Arms: Astegolimab SC Q2W; Astegolimab SC Q4W
Drug: Placebo — Participants will receive SC placebo Q2W
  Arms: Placebo SC Q2W

SUMMARY:
This study will evaluate the efficacy and safety of astegolimab compared with placebo in participants with chronic obstructive pulmonary disease (COPD) who are former or current smokers and have a history of frequent exacerbations.

ELIGIBILITY:
Inclusion Criteria

* Documented COPD diagnosis for ≥ 12 months
* History of frequent exacerbations, defined as having had 2 or more moderate or severe COPD exacerbations within 12 months prior to screening
* Post-bronchodilator FEV1 ≥ 20% and < 80% of predicted at screening
* Post-bronchodilator FEV1/FVC < 0.70 at screening
* Modified Medical Research Council (dyspnea scale) (mMRC) score ≥ 2
* Current tobacco smoker or former smoker with a history of smoking ≥ 10 pack-years
* On optimized COPD maintenance therapy as defined below for ≥ 12 months prior to screening, and stable on current therapy for at least 4 weeks prior to screening: Inhaled corticosteroid (ICS) plus long-acting beta-agonist (LABA), Long-acting muscarinic antagonist (LAMA) plus LABA, ICS plus LAMA plus LABA
* Chest X-ray or computed tomography (CT) scan within 6 months prior to screening or chest X-ray during the screening period that confirms the absence of clinically significant lung disease besides COPD

Exclusion Criteria

* Current documented diagnosis of asthma
* History of clinically significant pulmonary disease other than COPD
* Diagnosis of 1-antitrypsin deficiency
* History of long-term treatment with oxygen at > 4.0 liters/minute
* Lung volume reduction surgery or procedure within 12 months prior to screening
* Individuals participating in, or scheduled for, an intensive COPD rehabilitation program (participants who are in the maintenance phase of a rehabilitation program are eligible)
* History of lung transplant
* Any infection that resulted in hospital admission for ≥ 24 hours and/or treatment with oral, IV, or IM antibiotics within 4 weeks prior to or during screening
* Upper or lower respiratory tract infection within 4 weeks prior to or during screening
* Treatment with oral, IV, or IM corticosteroids within 4 weeks prior to initiation of study drug
* Initiation of or change in non-biologic immunomodulatory or immunosuppressive therapy within 3 months prior to screening
* Unstable cardiac disease, myocardial infarction, or New York Heart Association Class III or IV heart failure within 12 months prior to screening

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1290 (Estimated)
Dates: Start 2022-12-29 (Actual); Primary Completion 2025-06-24 (Actual); Study Completion 2027-09-24 (Estimated)

PRIMARY OUTCOMES:
Annualized rate of moderate and severe COPD exacerbations over the 52-week treatment period | 52 weeks

SECONDARY OUTCOMES:
Time to first moderate or severe COPD exacerbation during the 52-week treatment period | 52 weeks
Absolute change from baseline in health-related quality of life (HRQoL) at Week 52 as assessed through the St. George's Respiratory Questionnaire-COPD (SGRQ-C) total score | Week 52
Absolute change from baseline in post-bronchodilator forced expiratory volume (FEV1) at Week 52 | Week 52
Absolute change from baseline in the Evaluating Respiratory Symptoms in Chronic Obstructive Pulmonary Disease (E-RS:COPD) total score at Week 52 | Week 52
Proportion of participants with improvement in HRQoL at Week 52 | Week 52
Annualized rate of severe COPD exacerbations over the 52-week treatment period | 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (461):
- United States (80):
  - Pinnacle Research Group, Anniston, Alabama
  - AllerVie Clinical Research, Birmingham, Alabama
  - Synexus Clinical Research US, Inc. - Birmingham, Birmingham, Alabama
  - University of Alabama at Birmingham, Birmingham, Alabama
  - SEC Clinical Research LLC - Dothan 2 - ClinEdge - PPDS, Dothan, Alabama
  - Pulmonary Associates PA, Glendale, Arizona
  - Synexus Clinical Research US, Inc. - Phoenix West, Glendale, Arizona
  - AES - DRS - Synexus Clinical Research US, Inc. - Tucson, Tucson, Arizona
  - Lynn Institute of The Ozarks - ERN - PPDS, Little Rock, Arkansas
  - Kern Research, Bakersfield, California
  - VA Palo Alto Health Care System, Palo Alto, California
  - AES - DRS - Synexus Clinical Research US, Inc. - Vista, Vista, California
  - Allergy & Asthma Medical Group of the Bay Area, Walnut Creek, California
  - Cornerstone Research Institute, Altamonte Springs, Florida
  - Invictus Clinical Research Group, LLC, Coconut Creek, Florida
  - Finlay Medical Research Corporation, Greenacres City, Florida
  - San Marcus Research Clinic Inc., Miami, Florida
  - Oceane7 Medical & Research Center, Inc., Miami, Florida
  - Avantis Clinical Research, LLC, Miami, Florida
  - Research Institute of South Florida Inc, Miami, Florida
  - Diverse Clinical Research, LLC, Miami, Florida
  - Central Florida Pulmonary Group, PA, Orlando, Florida
  - Revival Clinical Research, Orlando, Florida
  - Florida Institute for Clinical Research, LLC, Orlando, Florida
  - Ormond Beach Clinical Research, Ormond Beach, Florida
  - Tampa Bay Health Care, Tampa, Florida
  - AES - DRS - Synexus Clinical Research US, Inc. - The Villages, The Villages, Florida
  - AES - DRS - Synexus Clinical Research US, Inc. - Atlanta, Atlanta, Georgia
  - Allergy Center at Brookstone Research - Centricity Research - HyperCore - PPD, Columbus, Georgia
  - Pivotal Research Solutions, Stonecrest, Georgia
  - ASHA Clinical Research - ClinEdge - PPDS, Hammond, Indiana
  - The Research Group of Lexington, LLC, Lexington, Kentucky
  - Best Clinical Trials, New Orleans, Louisiana
  - Paul A. Shapero, MD, PA, Bangor, Maine
  - Pulmonary Research Institute of Southeast Michigan, Farmington Hills, Michigan
  - Flushing Road Internal Medicine and Pediatrics - F, Flint, Michigan
  - Revive Research Institute, Lathrup Village, Michigan
  - Oakland Medical Research Center, Troy, Michigan
  - Washington University School of Medicine in St. Louis, St Louis, Missouri
  - Nebraska Medical Research Institute, Inc. - CRN, Bellevue, Nebraska
  - Machuca Family Medicine, Las Vegas, Nevada
  - Renown Regional Medical Center Hospital, Reno, Nevada
  - Hassman Research Institute - HRI - Berlin - CenExel - PPDS, Marlton, New Jersey
  - AES - DRS - Synexus Clinical Research US, Inc. - New York, New York, New York
  - WellNow Urgent Care and Clinical Research - Niskayuna, Schenectady, New York
  - Research Carolina Elite, Denver, North Carolina
  - Care Access Research - Fayetteville - PPDS, Fayetteville, North Carolina
  - Clinical Research of Gastonia, Gastonia, North Carolina
  - Pulmonix LLC, Greensboro, North Carolina
  - Advanced Respiratory and Sleep Medicine, PLLC, Huntersville, North Carolina
  - Southeastern Research Center, Winston-Salem, North Carolina
  - Wellnow Urgent Care and Research ? Springdale, Cincinnati, Ohio
  - WellNow Urgent Care & Research - Huber Heights, Huber Heights, Ohio
  - OK Clinical Research, Edmond, Oklahoma
  - Vital Prospects Clinical Research Institute PC - CRN, Tulsa, Oklahoma
  - The Oregon Clinic, Portland, Oregon
  - Clinical Research Associates Of Central Pa , Llc, Altoona, Pennsylvania
  - Allergy & Clinical Immun Assoc, Pittsburgh, Pennsylvania
  - Medtrial, LLC, Columbia, South Carolina
  - Velocity Clinical Research - Gaffney - PPDS, Gaffney, South Carolina
  - Care Access Research - Mauldin - PPDS, Mauldin, South Carolina
  - ClinSearch, LLC, Chattanooga, Tennessee
  - Clinical Trials Center of Middle Tennessee, Franklin, Tennessee
  - Tennessee Comprehensive Lung & Sleep Center, Hendersonville, Tennessee
  - FutureSearch Trials of Neurology, Austin, Texas
  - TTS Research, Boerne, Texas
  - Corsicana Medical Research, Corsicana, Texas
  - Baylor University Medical Center, Dallas, Texas
  - Epic Medical Research LLC - DeSoto, DeSoto, Texas
  - Greater Heights Memorial Pulmonary and Sleep, Houston, Texas
  - Trio Clinical Trials, Houston, Texas
  - Baylor College of Medicine Medical Center, Houston, Texas
  - Uni of Texas Health Science Center At Houston, Houston, Texas
  - Clinical Trial Network, Houston, Texas
  - Biopharma Informatic - Park Row - PPDS, Houston, Texas
  - Advances In Health Inc, Houston, Texas
  - R & H Clinical Research, Katy, Texas
  - University of Vermont Medical Center, Burlington, Vermont
  - Western Washington Medical Group, Everett, Washington
  - Allergy Asthma and Sinus Center-Greenfield, Greenfield, Wisconsin
- Argentina (22):
  - Consultorios Medicos Organizacion de Buen Ayre SRL, Buenos Aires
  - Nexo Salud Investigacion Clinica - Riobamba 429, Buenos Aires
  - CINME S.A. ? Centro de Investigaciones Metabolicas - Rx Trials LLC, Buenos Aires
  - Fundacion Faicep, Buenos Aires
  - Instituto de Investigaciones En Alergia Y Enfermedades Respiratorias, Buenos Aires
  - AES - AS - Glenny Corp. S.A. Buenos Aires, Buenos Aires
  - Centro de Medicina Respiratoria, Concepción del Uruguay
  - Sanatorio de la Canada, Córdoba
  - Framingham Centro Medico, La Plata
  - Centro Medico Capital, La Plata
  - Centro Platense en Investigaciones Respiratorias, La Plata
  - Centro Medico Dharma, Mendoza
  - Centro Privado de Medicina Respiratoria, Paraná
  - Sala de primeros auxilios Alberto Mignaburu, Ranelagh, Berazategui
  - Instituto Medico de la Fundacion Estudios Clinicos, Rosario
  - Servicio de Investigacion de Patologias Alergicas-Instituto ABC, Rosario
  - Sanatorio Parque de Rosario, Rosario
  - Centro Modelo de Cardiologia, San Miguel de Tucumán
  - Centro Medico San Nicolas Grupo Orono, San Nicolás de los Arroyos
  - CEPROSS- Centro Profesional San Salvador, San Salvador
  - Instituto Del Buen Aire, Santa Fe
  - Centro de Diagnostico Y Rehabilitacion, Santa Fe
- Institute for Respiratory Health - Midland, Midland, South Australia, Australia
- Austria (2):
  - Ordination Dr. Robert Voves, Feldbach
  - Ordination fur Lungenkrankheiten, Linz
- Belgium (4):
  - AZ Sint-Jan Brugge-Oostende, Bruges
  - Universitair Ziekenhuis Brussel, Brussels
  - Cliniques Universitaires Saint-Luc, Brussels
  - CHU de Liège, Liège
- Brazil (11):
  - CEDOES - Diagnóstico e Pesquisa, Vitória, Espírito Santo
  - L2IP ?Instituto de Pesquisas Clínicas Ltda., Brasília, Federal District
  - Santa Casa de Misericordia de Belo Horizonte - PPDS, Belo Horizonte, Minas Gerais
  - Instituto Méderi de Pesquisa e Saúde, Passo Fundo, Rio Grande do Sul
  - LMK Servicos Medicos SS, Porto Alegre, Rio Grande do Sul
  - Hospital Sao Lucas Da Pontificia Universidade Catolica Do Rio Grande Do Sul (PUCRS), Porto Alegre, Rio Grande do Sul
  - Universidade Estadual Paulista Julio de Mesquita Filho Faculdade de Medicina Campus de Botucatu, Botucatu, São Paulo
  - Faculdade de Medicina do ABC - FMABC, Santo André, São Paulo
  - CEMEC - Centro Multidisciplinar de Estudos Clínicos, São Bernardo do Campo, São Paulo
  - IBPCLIN Instituto Brasil de Pesquisa Clinica, Rio de Janeiro
  - Instituto do Coracao - HCFMUSP, São Paulo
- Bulgaria (15):
  - Multiprofile Hospital for Active Treatment Puls AD PPDS, Blagoevgrad
  - Multiprofile Hospital For Active Treatment Sveta Ekaterina - Dimitrovgrad EOOD, Dimitrovgrad
  - Multiprofile Hospital For Active Treatment Dr. Tota Venkova JSC, Gabrovo
  - Medical Center Hera EOOD, Montana
  - Multiprofile Hospital for Active Treatment Plovdiv, Plovdiv
  - Multiprofile Hospital for Active Treatment Sv. Ivan Rilski- Razgrad AD, Razgrad
  - Multiprofile Hospital for Active Treatment Shumen, Shumen
  - Multiprofile Hospital for Active Treatment - Silistra AD, Silistra
  - Multiprofile Hospital For Active Treatment - Dr. Bratan Shukerov AD, Smolyan
  - Fifth Multiprofile Hospital for Active Treatment - Sofia EAD, Sofia
  - Diagnostic-Consultative Center Aleksandrovska EOOD, Sofia
  - Diagnostic- Consultative Center Convex EOOD, Sofia
  - AES DRS Medical Center Synexus Sofia EOOD, Sofia
  - Diagnostic Consultative Centre Mladost?M OOD, Varna
  - Medical Center Tara OOD, Veliko Tarnovo
- Canada (11):
  - Edmonton Respiratory Consultants, Edmonton, Alberta
  - Office of Irvin Mayers, MD, Edmonton, Alberta
  - Synergy Respiratory & Cardiac Care - Synergy Wellness Centre Location, Sherwood Park, Alberta
  - Vancouver General Hospital, Vancouver, British Columbia
  - Dynamic Drug Advancement Ltd., Ajax, Ontario
  - Inspiration Research, Toronto, Ontario
  - Dr. Syed Anees Medicine Profession Corporation, Windsor, Ontario
  - Dr Anil Dhar Professional Medicine Corporation, Windsor, Ontario
  - Recherche GCP Research, Montreal, Quebec
  - Clinique de pneumologie et du sommeil de Lanaudiere, Saint-Charles-Borromée, Quebec
  - Centre Hospitalier de l'Universite Laval, Québec
- Chile (3):
  - Centro Respiratorio Integral LTDA. (CENRESIN), Pavie Gallegos
  - Oncocentro APYS, Viña del Mar
  - Fundacion Medica San Cristobal, Vitacura
- China (41):
  - The Third Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - Affiliated Hospital of Guangdong Medical University, Zhanjiang, Guangdong
  - Affiliated Hospital of Zunyi Medical University, Zunyi, Guizhou
  - The First People's Hospital of Lian Yun Gang, Lianyungang, Jiangsu
  - Beijing Chaoyang Hospital Capital Medical University, Beijing
  - China-Japan Friendship Hospital, Beijing
  - Beijing Jingmei Group General Hospital, Beijing
  - Peking University Third Hospital, Beijing
  - Beijing Hospital, Beijing
  - Peking University Shougang Hospital, Beijing
  - The First Hospital of Jilin University, Changchun
  - The First Hospital of Changsha, Changsha
  - The Third Hospital of Changsha, Changsha
  - West China Hospital, Sichuan University, Chengdu
  - Chengdu Fifth People's Hospital, Chengdu
  - The Southwest Hospital of Army Medical University, Chongqing
  - Army Medical Center of PLA(Daping Hospital), Chongqing
  - Guangzhou First People's Hospital, Guangzhou
  - Hainan General Hospital, Haikou
  - Hangzhou First People's Hospital, Hangzhou
  - Anhui Chest Hospital, Hefei
  - Huizhou Central People's Hospital, Huizhou
  - Taizhou Hospital of Zhejiang Province, Linhai
  - Jiangxi Provincial People's Hospital, Nanchang
  - Zhongda Hospital Southeast University, Nanjing
  - Nantong First People's Hospital, Nantong
  - Jiangxi Pingxiang People's Hospital, Pingxiang
  - Huadong Hospital Affiliated to Fudan University, Shanghai
  - Shengjing Hospital of China Medical University, Shenyang
  - Tianjin Medical University General Hospital, Tianjin
  - Central Hospital of Wuhan, Wuhan
  - Wuxi People's Hospital, Wuxi
  - Jiangyin People's Hospital, Wuxi
  - Xi'an International Medical Center Hospital, Xi'an
  - Zhongshan Hospital Xiamen University, Xiamen
  - Xinxiang First People's Hospital, Xinxiang
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou
  - Yangzhou First People?s Hospital, Yangzhou
  - The Fifth Affiliated Hospital Sun Yat-Sen University, Zhuhai
  - Zigong First People's Hospital, Zigong
- Czechia (9):
  - Plicní ambulance MUDr. I. Cierná Peterová s.r.o., Brandýs nad Labem-Stará Boleslav
  - Klinika nemoci plicnich a TBC FN Brno a LF MU - Ji, Brno
  - Fakultni nemocnice Hradec Kralove, Hradec Králové
  - Nemocnice Kyjov, prispevkova organizace, Kyjov
  - Odborna plicni ambulance Opava s.r.o, Opava
  - Ordinace chorob plicních s.r.o., Prague
  - AES - DRS - Synexus Czech s.r.o., Prague
  - Nemocnice Tabor, a.s., Tábor
  - Plicni stredisko Teplice s.r.o., Teplice
- Denmark (2):
  - Naestved Sygehus, Næstved
  - Sjaellands Universitetshospital, Roskilde, Roskilde
- France (5):
  - Sas Clinique De L Europe - Amiens, Amiens
  - Hopital Calmette, Lille
  - Groupe Hospitalier Cochin St Vincent de Paul La Roche Guyon, Paris
  - Hopital Haut Leveque, Pessac
  - CHU de Nancy-Hopital Brabois Adulte, Vandœuvre-lès-Nancy
- Germany (19):
  - Velocity Clinical Research Leipzig GmbH, Lübeck, Schleswig-Holstein
  - Praxis fur Kardiologie und Pneumologie Dr. med. Karin Forster, Berlin
  - Studienpraxis Berlin-Brandenburg, Berlin, Berlin
  - AES - DRS - Synexus Berlin Research Centre, Berlin
  - Lungenzentrum Darmstadt, Darmstadt
  - AES - DRS - Synexus Frankfurt Research Centre, Frankfurt
  - Universitaetsklinikum Frankfurt, Frankfurt
  - Clinical Research Hamburg, Hamburg
  - Praxisgem. Dres. Schmoller und Ehlers, Hamburg
  - Pneumologicum, Hanover
  - University Clinic Heidelberg, Heidelberg
  - Lungenfachklinik Immenhausen, Immenhausen
  - AES - DRS - Synexus Leipzig Research Centre, Leipzig
  - BAG Prof. Dr. G. Hoheisel Dr. A. Bonitz, Leipzig
  - SMO.MD GmbH, Magdeburg
  - Praxis Dr. med. Jan Feimer, München
  - Institut fur klinische Forschung GmbH, Neu-Isenburg
  - framol-med GmbH, Rheine
  - Klinikum Rosenheim, Rosenheim
- Greece (7):
  - University General Hospital of Alexandroupolis, Alexandroupoli
  - Evangelismos General Hospital of Athens, Athens
  - Navy Hospital of Athens, Athens
  - University General Hospital of Heraklion, Heraklio
  - University General Hospital of Ioannina, Ioannina
  - Iatriko Palaiou Falirou, Palaió Fáliro
  - Georgios Papanikolaou General Hospital of Thessaloniki, Thessaloniki
- Queen Mary Hospital, Hong Kong, Hong Kong
- Hungary (3):
  - Benyovszky Medical Center, Budapest
  - Omnimodus Elixír Kft., Csorna
  - Veszprem Megyei Tudogyogyintezet, Farkasgyepű
- India (15):
  - Paarthiv Lung Care Center, Hyderabad, Andhra Pradesh
  - Yashoda Hospitals Hitec City, Hyderabad, Andhra Pradesh
  - Government Medical College and Government General Hospital, Srikakulam, Andhra Pradesh
  - GMERS Medical College and Hospital, Sola, Ahmedabad, Gujarat
  - ESIC Medical College and Hospital - Faridabad, Faridabad, Haryana
  - Karnataka Medical College and Research Institute, Hubballi;Department of Medicine, Hubballi, Karnataka
  - Shree Hospital And Critical Care Centre, Nagpur, Maharashtra
  - Kothrud Hospital, Pune, Maharashtra
  - Aakash Healthcare Super Speciality Hospital, New Delhi, National Capital Territory of Delhi
  - Sawai Man Singh Hospital and Medical College, Jaipur, Rajasthan
  - Maharaja Agrasen Super Speciality Hospital, Jaipur, Rajasthan
  - Jawaharlal Nehru Medical College (JNMC), Aligarh, Uttar Pradesh
  - Apollo Spectra Hospital, Kanpur, Uttar Pradesh
  - MV Hospital and Research Centre, Lucknow, Uttar Pradesh
  - Institute of Post Graduate Medical Education and Research (IPGMER) and SSKM Hospital, Kolkata, West Bengal
- Israel (5):
  - Soroka University Medical Centre, Beersheba
  - Rambam Medical Center - PPDS, Haifa
  - Lady Davis Carmel Medical Center, Haifa
  - Hadassah Medical Center, Jerusalem
  - Meir Medical Center, Kfar Saba
- Italy (12):
  - Presidio Ospedaliero Santa Maria della Speranza, Battipaglia, Campania
  - Azienda Ospedaliera Dei Colli, Napoli, Campania
  - Azienda Ospedaliero-Universitaria di Ferrara - Arcispedale Sant' Anna, Ferrara, Emilia-Romagna
  - Arcispedale Santa Maria Nuova, Reggio Emilia, Emilia-Romagna
  - Fondazione PTV Policlinico Tor Vergata, Rome, Lazio
  - ASST Fatebenefratelli Sacco - Ospedale Luigi Sacco, Milan, Lombardy
  - Fondazione IRCCS Policlinico San Matteo di Pavia, Pavia, Lombardy
  - Azienda Sanitaria Ospedaliera S Luigi Gonzaga, Orbassano, Piedmont
  - Azienda Ospedaliero Universitaria Policlinico Vittorio Emanuele, Catania, Sicily
  - Azienda Ospedaliera Universitaria Policlinico Paolo Giaccone, Palermo, Sicily
  - Azienda Ospedaliera Universitaria Careggi, Florence, Tuscany
  - Azienda Ospedaliero Universitaria Senese - Policlinico Santa Maria alle Scotte, Siena, Tuscany
- Japan (61):
  - Makita Hospital, Sapporo, Hokkaido
  - Miura Medical Clinic, Miura-shi, Kanagawa
  - Yokohama Front Clinic, Yokohama, Kanagawa
  - Yokohama-Gumyouji Kokyuukinaika Naika Clinic, Yokohama, Kanagawa
  - Matsusaka City Hospital, Matsusaka-Shi, Mie-ken
  - University of the Ryukyus Hospital, Ginowan-shi, Okinawa
  - Fujieda Municipal General Hospital, Fujieda-Shi, Shizuoka
  - Yamaguchi University Hospital, Ube-shi, Yamaguchi
  - Asahikawa Medical Center, Asahikawa-shi
  - Fukuoka University Chikushi Hospital, Chikushino-shi
  - National Hospital Organization Kyushu Medical Center, Chuo-ku, Fukuoka-shi
  - Fukuwa Clinic, Chūōku
  - Fukuoka University Hospital, Fukuoka
  - Nishi Fukuoka Hospital, Fukuoka-Shi Nishi-Ku
  - Terada Respiratory and Internal Clinic, Himeji
  - Hiroshima Prefectural Hospital, Hiroshima
  - Ishikawa Prefectural Central Hospital, Ishikawa
  - National Hospital Organization Minami Kyoto Hospital, Jōyō
  - Kagoshima Kouseiren Hospital, Kagoshima
  - Kagoshima University Hospital, Kagoshima
  - Yokohama City University Medical Center, Kanagawa
  - Osaka-Minami Medical Center, Kawachinagano-Shi
  - Kiryu Kosei General Hospital, Kiryū
  - Kishiwada City Hospital, Kishiwada
  - Hospital of the University of Occupational and Environmental Health,Japan, Kitakyushu-shi
  - Juntendo Tokyo Koto Geriatric Medical Center, Kōtō City
  - Saiseikai Kumamoto Hospital, Kumamoto
  - Rakuwakai Otowa Hospital, Kyoto
  - National Hospital Organization Kyoto Medical Center, Kyoto
  - Machida Municipal Hospital, Machida-shi
  - Dokkyo Medical University Hospital, Mibu-Machi
  - Fukushima Medical University Hospital, Miyagi
  - Nagoya Ekisaikai Hospital, Nagoya
  - Kojunkai Social Medical Corporation Daido Clinic, Nagoya-shi Minami-ku
  - National Hospital Organization Ibarakihigashi National Hospital, Naka-gun
  - Niigata City General Hospital, Niigata
  - National Hospital Organization Okayama Medical Center, Okayama
  - Okayama Rosai Hospital, Okayama-Shi Minami-ku
  - Omuta National Hospital, Omuta
  - Izumi City General Hospital, Osaka
  - Oita Medical Center, Ōita
  - National Hospital Organization - Sagamihara National Hospital, Sagamihara-shi Minami-ku
  - Sakaide City Hospital, Sakaidechō
  - NHO Kinki-Chuo Chest Medical Center, Sakaishi
  - Japan Community Health Care Organization Hokkaido Hospital, Sapporo
  - Idaimae Minami 4-Jo Internal Medicine, Sapporo-shi Chuo-ku
  - Shizuoka City Shizuoka Hospital, Shizuoka
  - Iwata City Hospital, Shizuoka
  - Kamei Internal Medicine and Respiratory Clinic, Takamatsu
  - National Hospital Organization Takasaki General Medical Center, Takasaki
  - Minami Wakayama Medical Center, Tanabe
  - Tokyo-Eki Center-building Clinic, Tokyo
  - Nihon University Itabashi Hospital, Tokyo
  - Japanese Red Cross Medical Center, Tokyo
  - Toyama Prefectural Central Hospital, Toyama
  - Yamagata University Hospital, Yamagata
  - Nagata Hospital, Yanagawa
  - Showa University Fujigaoka Hospital, Yokohama-shi Aoba-ku
  - Kanagawa Cardiovascular and Respiratory Center, Yokohama-shi Kanazawa-ku
  - National Hospital Organization - Yokohama Medical Center, Yokohama-Shi Totsuka-Ku
  - Sanyudo Hospital, Yonezawa
- Kenya (6):
  - KEMRI-MTWAPA Clinical Trial Site, Kilifi, Coast
  - Clinical Research Health Network (CREA-N), Machakos
  - KEMRI CRDR Clinical Research Clinic Nairobi, Nairobi
  - University of Nairobi Clinical Research Centre, Nairobi
  - KEMRI/CRDR Siaya Clinical Research Annex, Siaya
  - Center for Research In Tropical Medicine and community development, Thika
- Latvia (6):
  - Health Center Association, Medical Center OLVI, Daugavpils
  - Daugavpils Regional Hospital, Daugavpils
  - Pauls Stradins Clinical University Hospital, R?ga
  - Riga 1st Hospital, Riga
  - ConsiliumMedicum, Riga
  - Postgraduate Medical Training Institute University of Latvia, Riga
- Netherlands (3):
  - Meander Medisch Centrum, Amersfoort
  - Martini Ziekenhuis, Groningen
  - Zuyderland Medisch Centrum - Heerlen, Heerlen
- New Zealand (5):
  - Greenlane Clinical Centre, Auckland
  - Dunedin Hospital, Dunedin
  - Waikato Hospital, Hamilton
  - P3 Research, Tauranga
  - P3 Research - Kapiti - PPDS, Waikanae Beach
- Philippines (7):
  - Manila Central University-Filemon D Tanchoco Medical Foundation, Caloocan
  - CARE CT Group Inc., Dasmariñas
  - Healthlink Medicalsurgicaldental Clinic and Diagnostic Center, Iloilo City
  - West Visayas State University Medical Center, Iloilo City
  - Mary Mediatrix Medical Center, Lipa City
  - Philippine Heart Center, Quezon City
  - Quirino Memorial Medical Center, Quezon City
- Poland (29):
  - CenterMed Sp. z o.o., Tarnów, Lesser Poland Voivodeship
  - AppleTreeClinics Network Sp. z o.o., Lodz, Lódzkie
  - Centrum Medycyny Oddechowej Mroz sp. j., Bia?ystok
  - Vitamed Galaj i Cichomski sp.j., Bydgoszcz
  - Medical Center Kermed, Bydgoszcz
  - Centrum Medyczne Lukamed Joanna Luka-Wendrowska, Chojnice
  - AES - DRS - Synexus Polska Sp. z o.o. Oddzial w Czestochowie, Częstochowa
  - AES - DRS - Synexus Polska Sp. z o.o. Oddzial w Gdansku, Gda?sk
  - Synexus Polska Sp. z o.o. Oddzial w Gdyni, Gdynia
  - Centrum Medyczne CLW-med Aneta Cichomska , Joanna Luka -Wendrowska, Grudzadz
  - Prywatny Gabinet Pulmonologiczny Joanna Nowacka-Apiyo, Grudziądz
  - Centrum Medyczne Katowice - PRATIA - PPDS, Katowice
  - Wojewodzki Szpital Specjalistyczny im. Ludwika Rydygiera w Krakowie, Krakow
  - Prywatna Praktyka Lekarska Adam Smialowski, Ksawerów
  - AES - DRS - Synexus Polska Sp. Z o.o. Oddzial w Lodzi, Lodz
  - Clinical Best Solutions - Lublin, Lublin
  - NZOZ Przychodnia Alergologiczno-pulmonologiczna, Lublin
  - ABC-Pulmo NZOZ Agnieszka Dobielska, Jaroslaw Dobie, Radom
  - Centrum Medyczne KARDIOTEL, Sopot
  - Kiepury Clinic, Sosnowiec
  - Gabinet Pulmonologii i Diagnostyki Chorob Alergicznych Dorota Malosek, Szczecin
  - NZOZ Poradnia Chorob Pluc i Alergologii, Słupsk
  - MICS Centrum Medyczne Torun, Torun
  - Viltis Medica Specjalistyczna Praktyka Lekarska Lek. Med. Agata Kot, Trzebnica
  - AES - DRS - Synexus Polska Sp. z o.o. Oddzial w Warszawie, Warsaw
  - Synexus Polska Sp. z o.o. Oddzial we Wroclawiu, Wroc?aw
  - Centrum Badan Klinicznych Piotr Napora Lekarze Spolka Partnerska, Wroc?aw
  - Lekarze Specjalisci J. Malolepszy i Partnerzy, Wroc?aw
  - Medical Center Clinhouse, Zabrze
- Allianze Pulmonary Research LLC, Guaynabo, Puerto Rico
- Romania (2):
  - Cardos Rosca Medical S.R.L., Cluj-Napoca
  - Fundatia CardioPrevent, Timișoara
- South Africa (10):
  - Iatros International, Bloemfontein, Free State
  - Newtown Clinical Research Centre, City of Johannesburg, Gauteng
  - Johese Clinical Research, Centurion
  - Dr. Ismail Abdullah Private Practice, City of Cape Town
  - CLINRESCO, ARWYP Medical Suites, Kempton Park
  - Ubuntu Clinical Research Sites, Krugersdorp
  - AES - DRS - Synexus Watermeyer Clinical Research Centre, Pretoria
  - Medicross Pretoria West, Jongaie Research, Pretoria
  - AES - DRS - Synexus - Helderberg Clinical Research Centre, Somerset West
  - Dr Yacoob AK Private Practice, Welkom
- South Korea (10):
  - Soon Chun Hyang University Hospital Bucheon, Bucheon-si
  - Chungbuk National University Hospital, Cheongju-si
  - Yeungnam University Hospital, Daegu
  - CHA Bundang Medical Center, Gyeonggi-do
  - Kangbuk Samsung Hospital, Seoul
  - Asan Medical Center - PPDS, Seoul
  - Samsung Medical Center - PPDS, Seoul
  - Chung-Ang University Hospital, Seoul
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul
  - Yonsei University Wonju Severance Christian Hospital, Wŏnju
- Spain (11):
  - Hospital Universitario Son Espases, Palma de Mallorca, Balearic Islands
  - Hospital El Bierzo, Ponferrada, LEON
  - Hospital Universitario de Torrejon, Torrejón de Ardoz, Madrid
  - Vithas Xanit International Hospital, Benalmádena Costa, Malaga
  - Hospital del Mar, Barcelona
  - Hospital Universitario La Paz - PPDS, Barcelona
  - Hospital Universitario de La Princesa, Madrid
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Clinico Universitario de Valencia, Valencia
  - Consorcio Hospital General Universitario de Valencia, Valencia
  - Hospital de La Ribera, Valencia
- Sweden (6):
  - Clinical Trial Consultants - Linkoping, Uppsala, Uppsala County
  - Sahlgrenska Universitetssjukhuset, Gothenburg
  - Universitetssjukhuset Orebro (USO), Örebro
  - Clinical Trial Consultants - Karolinska, Solna
  - Akardo AB, Stockholm
  - Clinical Trial Consultants - Uppsala, Uppsala
- Zurcher Reha Zentren Wald, Zurich, Switzerland
- Taiwan (7):
  - Changhua Christian Hospital, Chang-hua
  - Kaohsiung Medical University Hospital, Kaoshiung City
  - Far East Memorial Hospital, New Taipei City
  - Taipei Medical University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Tri-Service General Hospital, Taipei
  - Chang Gung Memorial Hospital - Linkou, Taoyuan District
- Thailand (3):
  - Chulalongkorn University, Bangkok
  - Srinagarind Hospital, Khon Kaen University, Khon Kaen
  - Central Chest Institute of Thailand, Muang
- Turkey (Türkiye) (6):
  - Sureyyapasa Gogus Hastaliklari ve Gogus Cerrahisi Egitim ve Arastirma Hastanesi, Istanbul
  - Kocaeli University Hospital, Kocaeli
  - Kirikkale Universitesi Tip Fakultesi Hastanesi, Kırıkkale
  - Mersin University Medical Faculty, Mersin
  - Rize Recep Tayyip Erdogan University Training and Research Hospital, Rize Merkez
  - Cukurova Universitesi Tip Fakultesi Balcali Hastanesi, Sarıçam
- United Kingdom (19):
  - Castle Hill Hospital, Cottingham, Yorkshire
  - AES - DRS - Synexus Scotland Clinical Research Centre, Bellshill
  - AES - DRS - Synexus Midlands Clinical Research Centre, Birmingham
  - AES - DRS - Synexus Wales Clinical Research Centre, Cardiff
  - Royal Primary Care - Ashgate Manor, Chesterfield
  - AES - DRS - NW Consortium Lancashire, Chorley
  - Lakeside Surgery, Corby
  - University Hospital Coventry, Coventry
  - Royal Infirmary of Edinburgh, Edinburgh
  - AES - DRS - Synexus Hexham Clinical Research Centre, Hexham
  - Velocity Clinical Research - High Wycombe - PPDS, High Wycombe
  - Royal Lancaster Infirmary, Lancaster
  - St James University Hospital, Leeds
  - Glenfield Hospital, Leicester
  - AES - DRS - NW Consortium Merseyside, Liverpool
  - Velocity Clinical Research North London - Percy Road - PPDS, London
  - St Thomas' Hospital, London
  - AES - DRS - NW Consortium Manchester, Manchester
  - Norfolk and Norwich University Hospital, Norwich

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing